CLINICAL TRIAL: NCT02268864
Title: A Phase 2, Open-label Study to Investigate the Efficacy and Safety of the Combination of Simeprevir and Daclatasvir in Chronic Hepatitis C Genotype 1b-Infected Subjects
Brief Title: A Study to Assess the Efficacy and Safety of the Combination of Simeprevir and Daclatasvir in Chronic Hepatitis C Genotype 1b-Infected Participants
Acronym: COMMIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR105490; 2014-003413-28 (EudraCT Number); TMC435HPC2019 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C Chronic; Simeprevir; Daclatasvir
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Simeprevir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simeprevir + Daclatasvir (Experimental): Participants who have Hepatitis C virus (HCV) genotype 1b infection with advanced fibrosis or compensated cirrhosis (METAVIR F3/F4) will receive simeprevir 150 milligram (mg) capsule and daclatasvir 60 mg tablet orally once daily for 12 or 24 weeks.
  Interventions: Drug: Simeprevir; Drug: Daclatasvir

INTERVENTIONS:
Drug: Simeprevir — Simeprevir 150 mg oral capsule will be administered once daily for 12 or 24 weeks.
Drug: Daclatasvir — Daclatasvir 60 mg oral tablet will be administered once daily for 12 or 24 weeks.

SUMMARY:
The purpose of this study is to determine the efficacy of a 12- or 24-week treatment regimen of simeprevir in combination with daclatasvir, as measured by sustain virologic response 12 (SVR12), in treatment-naive, chronic hepatitis C virus (HCV) genotype 1b-infected participants who have advanced fibrosis or compensated cirrhosis (METAVIR F3/F4).

DETAILED DESCRIPTION:
This is an open-label (all people know which treatment the participants receive) study to investigate the efficacy, safety and tolerability of simeprevir and daclatasvir in chronic Hepatitis (inflammation of the liver) C virus (HCV) genotype 1b infected participants who are treatment-naive. The total study duration for each participant will be approximately 40 weeks or approximately 52 weeks. The study will consist of 4 parts: Screening Phase (approximately 4 weeks) and open-label treatment Phase (12 weeks), optional open label treatment phase extension (12 Weeks) and follow-up Phase (up to Week 40 or Week 52). Participants will receive simeprevir (150 milligram [mg] capsule) and daclatasvir (60 mg tablet) orally once daily for 12 or 24 weeks. Efficacy will be primarily evaluated by percentage of participants with SVR12. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have chronic Hepatitis C virus (HCV) genotype 1b infection confirmed at Screening
* Participant must have HCV ribonucleic acid (RNA) greater than (>) 10,000 international unit per milliliter (IU/mL) at Screening
* Participant must have documented fibrosis stage at Screening (or between Screening and Day 1 [baseline]). Liver disease will be staged based on one of the following methods. a) Shear wave elastography (Fibroscan) within less than or equal to (<=) 6 months before Screening or between Screening and Day 1 (baseline). METAVIR F3 > 9.6 Kilopascals (kPa) and the cut-off for cirrhosis is greater than or equal to (>=) 14.6 kPa. b) A biopsy documenting METAVIR F3-F4. Biopsy performed within the 24 months before Screening will be accepted for participants with METAVIR score F3. For cirrhotic participants (METAVIR score F4) a biopsy performed at any previous time is acceptable
* Participants who have cirrhosis must have an hepatic imaging procedure (ultrasound, computed tomography [CT] scan or magnetic resonance imaging [MRI]) within 6 months prior to the Screening visit (or between Screening and Day 1) with no findings suspicious for hepatocellular carcinoma
* Participant must have a body mass index (BMI) >= 18 Kilogram per meter^2 (kg/m^2)
* Participant must be treatment naive (that is, have not received prior treatment for HCV with any approved or investigational drug)

Exclusion Criteria:

* Participant has co-infection with HCV of another genotype; a) Participant who has HCV genotype 1b has coinfection with HCV of a genotype other than genotype 1b
* Chronic HCV genotype 1b-infected participant who has the presence of genetic variants coding for the NS5A-Y93H and/or L31M/V amino acid substitutions at Screening
* Participant has evidence of current or previous episodes of hepatic decompensation (including controlled or uncontrolled ascites, bleeding varices or hepatic encephalopathy)
* Participant has chronic liver disease of a non-HCV etiology (including but not limited to hemochromatosis, Wilson's disease, alfa 1-antitrypsin deficiency, cholangitis, drug- or alcohol-related liver disease, primary biliary cirrhosis)
* Participant has any other uncontrolled clinically significant disease or clinically significant findings during Screening that in the opinion of the investigator could compromise the participants' safety or could interfere with the participant participating in and completing the study
* Participant has coinfection with hepatitis A or hepatitis B virus (hepatitis A antibody immunoglobulin M [IgM] or hepatitis B surface antigen [HBsAg] positive at Screening)
* Participant has received a solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (23):
- Belgium (3):
  - Antwerp
  - Brussels
  - Ghent
- France (6):
  - Créteil
  - Lyon
  - Montpellier
  - Nice
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Frankfurt
  - Hamburg
  - Hanover
  - Kiel
  - Tübingen
  - Würzburg
- Hungary (2):
  - Budapest
  - Debrecen
- Spain (4):
  - Badalona
  - Barcelona
  - Santander
  - Valencia
- United Kingdom (2):
  - Birmingham
  - London

REFERENCES:
- [Derived] Hezode C, Almasio PL, Bourgeois S, Buggisch P, Brown A, Diago M, Horsmans Y, Serfaty L, Szalay F, Gaeta GB, Planas R, Schlag M, Lonjon-Domanec I, Omoruyi E, DeMasi R, Zeuzem S. Simeprevir and daclatasvir for 12 or 24 weeks in treatment-naive patients with hepatitis C virus genotype 1b and advanced liver disease. Liver Int. 2017 Sep;37(9):1304-1313. doi: 10.1111/liv.13376. Epub 2017 Mar 13. PMID 28135777

RESULTS

PARTICIPANT FLOW:
Groups:
- 12 Weeks Prior Amendment: Simeprevir 150 milligram (mg) once daily as an oral capsule in combination with daclatasvir 60 mg once daily as an oral tablet for participants who completed the 12-week treatment before Amendment 3 of the protocol was implemented.
- 12 Weeks Post Amendment: Simeprevir 150 mg once daily as an oral capsule in combination with daclatasvir 60 mg once daily as an oral tablet for participants who opted for a 12-week treatment period after amendment.
- 24 Weeks Extension: Simeprevir 150 mg once daily as an oral capsule in combination with daclatasvir 60 mg once daily as an oral tablet for participants who opted for an extended 24-week treatment after amendment.
Period: Overall Study
Arm/Group | 12 Weeks Prior Amendment | 12 Weeks Post Amendment | 24 Weeks Extension
Started | 17 | 25 | 64
Completed | 15 | 24 | 64
Not Completed | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set is defined as all participants who received at least one dose of simeprevir or daclatasvir.
Groups:
- Total: Total of all reporting groups
Arm/Group | 12 Weeks Prior Amendment | 12 Weeks Post Amendment | 24 Weeks Extension | Total
Number analyzed (Participants) | 17 | 25 | 64 | 106
Age, Continuous [Median (Full Range); unit: years] | 53.0 (15.34) [21 to 82] | 64.0 (14.77) [25 to 83] | 59.0 (12.6) [26 to 83] | 59.0 (13.53) [21 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 27 | 43
  Male | 12 | 14 | 37 | 63
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 6 | 1 | 5 | 12
  France | 3 | 3 | 19 | 25
  Germany | 3 | 3 | 14 | 20
  Hungary | 4 | 0 | 8 | 12
  Italy | 0 | 10 | 6 | 16
  Spain | 1 | 8 | 11 | 20
  United Kingdom | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After End of Study Drug Treatment (SVR12)
Description: Participants were considered to have reached SVR12, if 12 weeks after the actual end of treatment (EOT), hepatitis C virus (HCV) ribonucleic acid (RNA) was less than lower limit of quantification (<LLOQ) (detectable or undetectable).
Time Frame: At 12 weeks after end of treatment
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 Weeks Prior Amendment | 12 Weeks Post Amendment | 24 Weeks Extension
Number analyzed (Participants) | 17 | 25 | 64
percentage of participants | 70.6 [44.04 to 89.69] | 100 [86.28 to 100] | 93.8 [84.76 to 98.27]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After End of Study Drug Treatment (SVR4)
Description: Participants were considered to have reached SVR4, if 4 weeks after the actual EOT, HCV RNA was <LLOQ (detectable or undetectable).
Time Frame: At 4 weeks after actual EOT
Population: The ITT analysis set is defined as all participants who received at least one dose of simeprevir or daclatasvir.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 Weeks Prior Amendment | 12 Weeks Post Amendment | 24 Weeks Extension
Number analyzed (Participants) | 17 | 25 | 64
percentage of participants | 70.6 [44.04 to 89.69] | 100 [86.28 to 100] | 93.8 [84.76 to 98.27]

3. Secondary Outcome: Percentage of Participants With SVR 24 Weeks After End of Study Drug Treatment (SVR 24)
Description: Participants were considered to have reached SVR24, if 24 weeks after the actual EOT, HCV RNA was <LLOQ (detectable or undetectable).
Time Frame: At 24 weeks after actual EOT
Population: The ITT analysis set is defined as all participants who received at least one dose of simeprevir or daclatasvir.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 Weeks Prior Amendment | 12 Weeks Post Amendment | 24 Weeks Extension
Number analyzed (Participants) | 17 | 25 | 64
percentage of participants | 70.6 [44.04 to 89.69] | 100 [86.28 to 100] | 93.8 [84.76 to 98.27]

4. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: Participants were considered on-treatment failures if they did not achieve SVR12 and had (confirmed) detectable HCV RNA, ie, <LLOQ detectable or greater than equal to (>=) LLOQ at EOT.
Time Frame: Up to Week 24 after actual EOT
Population: The ITT analysis set is defined as all participants who received at least one dose of simeprevir or daclatasvir.
Measure: Number; unit: percentage of participants
Arm/Group | 12 Weeks Prior Amendment | 12 Weeks Post Amendment | 24 Weeks Extension
Number analyzed (Participants) | 17 | 25 | 64
percentage of participants | 29.4 | 0.0 | 4.7

5. Secondary Outcome: Number of Participants With Viral Breakthrough
Description: Participants were considered to have had viral breakthrough if they had a confirmed greater than (>) 1.0 log10 international units/milliliter (IU/mL) increase in HCV RNA from nadir OR confirmed HCV RNA >100 IU/mL while previously having achieved HCV RNA <LLOQ when on study treatment.
Time Frame: Up to Week 24
Population: The ITT analysis set is defined as all participants who received at least one dose of simeprevir or daclatasvir.
Measure: Number; unit: participants
Groups:
- 12 Weeks Prior Amendment: Simeprevir 150 mg once daily as an oral capsule in combination with daclatasvir 60 mg once daily as an oral tablet for participants who completed the 12 week treatment before Amendment 3 of the protocol was implemented.
- 12 Weeks Post Amendment: Simeprevir 150 mg once daily as an oral capsule in combination with daclatasvir 60 mg once daily as an oral tablet for participants who opted for a 12 week treatment period after amendment.
- 24 Weeks Extension: Simeprevir 150 mg once daily as an oral capsule in combination with daclatasvir 60 mg once daily as an oral tablet for participants who opted for an extended 24 week treatment after amendment.
Arm/Group | 12 Weeks Prior Amendment | 12 Weeks Post Amendment | 24 Weeks Extension
Number analyzed (Participants) | 17 | 25 | 64
participants | 4 | 0 | 3

6. Secondary Outcome: Number of Participants With Viral Relapse
Description: Participants were considered to have had viral relapse if they did not achieve SVR12 and met the following conditions: had HCV RNA <LLOQ (undetectable) at EOT and had HCV RNA >=LLOQ during the follow-up period.
Time Frame: Up to Week 24 after actual EOT
Population: The ITT analysis set is defined as all participants who received at least one dose of simeprevir or daclatasvir.
Measure: Number; unit: participants
Arm/Group | 12 Weeks Prior Amendment | 12 Weeks Post Amendment | 24 Weeks Extension
Number analyzed (Participants) | 17 | 25 | 64
participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: Total number of participants at risk reported in the 12-24 weeks were the same participants who continued the 24-weeks extension period after completion of 1-12 weeks treatment phase (up to Day 88).
Groups:
- 1-12 Weeks: Simeprevir 150 mg once daily as an oral capsule in combination with Daclatasvir 60 mg once daily as an oral tablet for participants who has adverse events (AEs) that started before or on day 88 on treatment.
- 12-24 Weeks: Simeprevir 150 mg once daily as an oral capsule in combination with Daclatasvir 60 mg once daily as an oral tablet for participants who has AEs that started after day 88 on treatment.
Arm/Group | 1-12 Weeks | 12-24 Weeks
Serious Adverse Events (participants affected / at risk) | 4/106 | 3/64
Other Adverse Events (participants affected / at risk) | 44/106 | 2/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1-12 Weeks (N=106) | 12-24 Weeks (N=64)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Wound Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1-12 Weeks (N=106) | 12-24 Weeks (N=64)
Asthenia (General disorders) | 14 | 1
Fatigue (General disorders) | 16 | 1
Headache (Nervous system disorders) | 16 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.